CLINICAL TRIAL: NCT04325386
Title: Clozapine CHAMPION-ECHO (Center for Help and Assistance for Maryland Prescribers- Improving Outcomes Network Using Extension for Community Healthcare Outcomes); Randomized Educational Study to Improve Clozapine Prescribing Through a Project ECHO Model
Brief Title: Clozapine CHAMPION-ECHO Educational Study to Improve Clozapine Use.
Acronym: CHAMPION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Deanna Kelly, Cheif Treatment Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HP-00087399
Record Dates: First submitted 2020-02-11; First posted 2020-03-27 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia Schizoaffective
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: The investigators will compare an educational intervention between prescribers who individually enrolled from participating clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECHO Intervention (Experimental): Project ECHO (Extension for Community Healthcare Outcomes) based intervention 26 CME educational sessions. The sessions will include: 1) active dissemination of knowledge and information by an expert followed by 2) clozapine case presentations and vignettes. 1.25 hour long. Also consultation line and ATHELAS device.
  Interventions: Other: ECHO Intervention
- eTAU (Placebo Comparator): Consultation line and ATHELAS Device only
  Interventions: Other: eTAU

INTERVENTIONS:
Other: ECHO Intervention — Project ECHO (Extension for Community Healthcare Outcomes) based intervention 26 CME educational sessions. The sessions will include: 1) active dissemination of knowledge and information by an expert followed by 2) clozapine case presentations and vignettes. 1.25 hour long. Also consultation line and ATHELAS device.
  Arms: ECHO Intervention
Other: eTAU — Consultation Line and ATHELAS device only
  Arms: eTAU

SUMMARY:
In a randomized controlled design with approximately 26 biweekly sessions over 12 months, the investigators propose to test the effectiveness of an ECHO-based intervention for improving the use of clozapine in people eligible for clozapine. The sessions will include: 1) active dissemination of knowledge and information by an expert "hub" followed by 2) clozapine case presentations and vignettes submitted by the "spokes".

This intervention, Clozapine CHAMPION-ECHO (Center for Help and Assistance for Maryland Prescribers- Improving Outcomes Network using Extension for Community Healthcare Outcomes, will be referred to as "CHAMPION" throughout.. To minimize ANC monitoring barriers and maximize recruitment, the investigators will provide Food and Drug Administration (FDA)-cleared ANC point of care (POC) monitoring devices to all study sites, including those in the control condition. The investigators will enroll at least 300 prescribers and additional clinical team members (up to 300) from up to 60 mental health clinics (MHCs) and other treatment sites; approximately half the participants will be randomized to CHAMPION and half randomized to enhanced treatment as usual (ETAU).

ELIGIBILITY:
Inclusion Criteria:

* Located at a site in the State of Maryland with at least 3 prescribers at the site.
* Prescribers/clinical team should be licensed in the State of Maryland and have prescribed antipsychotics previously.
* Between the ages of 22 and 85 years old
* Willing to participate in pre- and post-testing
* Willing to agree to try to participate in the CHAMPION sessions

Exclusion Criteria:

* Not willing to participate in CHAMPION Sessions

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2024-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Psychiatric Research Center (MPRC) Treatment Research Program (TRP), Catonsville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As per grant and protocol all outcomes are by participant level no analysis by site.
Units Other Than Participants: Clinics
Groups:
- ECHO Intervention: Project ECHO (Extension for Community Healthcare Outcomes) based intervention sessions for improving the use of clozapine in people with treatment-resistant schizophrenia. The sessions will include: 1) active dissemination of knowledge and information by an expert followed by 2) clozapine case presentations and vignettes.
  Education Sessions: Project ECHO (Extension for Community Healthcare Outcomes) based intervention sessions for improving the use of clozapine in people with treatment-resistant schizophrenia. The sessions will include: 1) active dissemination of knowledge and information by an expert followed by 2) clozapine case presentations and vignettes.
- Enhanced Treatment As Usual (eTAU): No Education Session: No Education Session
Period: Overall Study
Arm/Group | ECHO Intervention | Enhanced Treatment As Usual (eTAU)
Started (Participants) | 126; 21 Clinics | 140; 22 Clinics
Completed (Participants) | 126; 21 Clinics | 140; 22 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Groups:
- Education Sessions: Project ECHO (Extension for Community Healthcare Outcomes) based intervention sessions for improving the use of clozapine in people with treatment-resistant schizophrenia. The sessions will include: 1) active dissemination of knowledge and information by an expert followed by 2) clozapine case presentations and vignettes.
  Education Sessions: Project ECHO (Extension for Community Healthcare Outcomes) based intervention sessions for improving the use of clozapine in people with treatment-resistant schizophrenia. The sessions will include: 1) active dissemination of knowledge and information by an expert followed by 2) clozapine case presentations and vignettes.
- No Education Sessions: No Education Session: No Education Session
- Total: Total of all reporting groups
Arm/Group | Education Sessions | No Education Sessions | Total
Number analyzed (Participants) | 126 | 140 | 266
Age, Customized [Count of Participants; unit: Participants]
  39 year or less | 47 | 58 | 105
  40-49 years | 39 | 33 | 72
  50-59 years | 16 | 33 | 49
  60 years or more | 24 | 16 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 100 | 193
  Male | 33 | 40 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 71 | 79 | 150
  Black | 32 | 32 | 64
  Other | 20 | 27 | 47
  Unknown | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 126 | 140 | 266

OUTCOME MEASURES:

1. Primary Outcome: Change in Clozapine Prescriptions Using Medicaid Claims Data
Description: The data outcome is new clozapine prescriptions by provider based on a variable linking provider ID to percent of clozapine prescriptions.
Time Frame: Baseline and endpoint changes after 12 month intervention
Measure: Mean (Standard Error); unit: Mean percent of Clozapine prescriptions
Groups:
- eTAU: No Education Session. Consultation Line and ATHELAS Device only
Arm/Group | ECHO Intervention | eTAU
Number analyzed (Participants) | 126 | 140
Mean percent of Clozapine prescriptions
  Mean percent of Clozapine prescriptions among antipsychotic prescribing Pre Intervention | 9.4 (0.70) | 10.8 (0.79)
  Mean percent of Clozapine prescriptions among antipsychotic prescribing Post intervention | 11.8 (0.92) | 9.5 (0.90)

2. Primary Outcome: Change in Prescriber Knowledge of Clozapine Use
Description: A 52 item Multiple Choice Questionnaire will be used to assess knowledge. The knowledge-based test questions will consist of 2 questions per 26 topic areas and will conform to best practices and guidelines for design of the questions. The total mean score will range from 0-52 with higher scores being better outcome. The questions were developed and validated by the team.
Time Frame: Baseline and endpoint changes after 12 month intervention
Measure: Mean (Standard Deviation); unit: Percentage of Correct responses reported
Groups:
- eTAU: No Education Session, Consultation Line and ATHELAS Device only
Arm/Group | Echo Intervention | eTAU
Number analyzed (Participants) | 126 | 140
Percentage of Correct responses reported
  Pre Intervention | 63 (12) | 66 (11)
  Post Intervention | 71 (17) | 67 (12)

3. Primary Outcome: Change in Self-reported Competence for Clozapine Use
Description: We will use a mean score on a Visual Analog Scale (VAS) (0-100 mm) for overall competence with higher scores being better outcome.
Time Frame: Baseline and endpoint changes after 12 month intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- eTAU: No Education Sessions. Consultation Line and ATHELAS Device only.
Arm/Group | ECHO Intervention | eTAU
Number analyzed (Participants) | 126 | 140
score on a scale
  Pre Sessions | 55.3 (21.0) | 59.0 (20.5)
  Post Sessions | 68.4 (22.3) | 71.4 (19.2)

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored or assessed
Description: Adverse Events were not monitored or assessed
Arm/Group | Education Sessions | No Education Sessions
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT04325386/Prot_SAP_000.pdf